CLINICAL TRIAL: NCT01429545
Title: Phase 2 Study of Clinical Utility of Combination Tocolysis in Preterm Labor
Brief Title: Single Versus Combination Therapy in Acute Tocolysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tawam Hospital (Other)
Responsible Party: Principal Investigator, Wafa Al Omari, Consultant Obstetrics and gynecolgy, Tawam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/95
Record Dates: First submitted 2011-09-01; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Preterm Labour
Keywords: Tocolysis; atosiban; nifedipine; combination
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — atosiban; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Atosiban (Active Comparator): Patients on single agent atosiban alone
  Interventions: Drug: Atosiban
- Group 2 (Experimental): Patients on combination of atosiban and nifedipine
  Interventions: Drug: Atosiban and nifedipine

INTERVENTIONS:
Drug: Atosiban — Atosiban was given as a bolus (6.7 mg. IV) over 1 min then an infusion of 18 mg/hr for 3 hrs followed by 6 mg/hr for 48 hrs.
  Other Names: Tractocile
  Arms: Group 1 - Atosiban
Drug: Atosiban and nifedipine — This group were given simultaneously as follows:Atosiban was given as a bolus (6.7 mg. IV) over 1 min then an infusion of 18 mg/hr for 3 hrs followed by 6 mg/hr for 48 hrs.Nifedipine was given in the dose of 10 mg orally every 15 min till uterine quiescence was achieved (<4 contractions/hr). Maximum dose was 40 mg in the first hour then maintenance dose of 10 mg every 4-6 h for 48 hrs was given.
  Other Names: Tractocile and nifedipine
  Arms: Group 2

SUMMARY:
The purpose of this study is to compare the tocolytic efficacy, effectiveness and safety of Atosiban in comparison with the combination of Atosiban and Nifedipine together.

DETAILED DESCRIPTION:
Preterm birth, defined as birth at less than 37+0 weeks of gestation, is the most important determinant of adverse infant outcomes. It accounts for 5 to 11% of births in the world, but represents the single largest cause of mortality and morbidity for newborns and a major cause of morbidity for pregnant women. These babies are at increased risk of cerebral palsies, chronic pulmonary insufficiency and other handicaps resulting in suboptimal performance in school and decreased abstractive thinking compared with infants born at term. The economic burden on society in catering for these preterm babies is high. A multi-level modeling of hospital service utilization and cost profile of preterm birth done in 2005 in the United Kingdom, has outlined the huge economic consequences of preterm birth in the first 10 years of life. Furthermore, recent data from Denmark have shown an overall increase in the proportion of preterm deliveries by 22% from 1995 to 2004(from 5.2% to 6.3%). Neonatal mortality has declined, mostly due to improved management of very low birth weight babies rather than prevention of preterm labor (PTL).

The most common treatment used in the management of PTL involves pharmacological inhibition of preterm uterine contractions. Perinatal death and morbidity resulting from PTL are not only strongly related to early gestational age but also to antenatal administration of steroids and transfer to a tertiary care centre in utero or after birth.6 Hence, the choice of tocolytic agent depends on its ability to delay the delivery by at least 48 hours from the time of administration of steroids and preferably longer without maternal or fetal side effects. There is considerable variation in the type of tocolytic agent used in different parts of the world. Single agent tocolysis using ritodrine (β-agonist), atosiban (oxytocin antagonist) or nifedipine (calcium channel blocker) is a common practice. Atosiban has been shown to have comparable effectiveness to β-agonists but with improved side-effect profile similar to that seen in placebo studies. Meta analysis from Cochrane systematic review failed to demonstrate the superiority of atosiban over betamimetics or placebo in terms of tocolytic efficacy or infant outcomes, but, the maternal drug reactions that required treatment cessation were fewer with atosiban. Nifedipine is the only agent associated with improved perinatal outcomes and fewer maternal side-effects than betamimetics. A direct comparison between atosiban and nifedipine has shown that both drugs are equally effective in acute tocolysis, however maternal side-effects were more pronounced with nifedipine.

Due to the differences in their pharmacokinetics and pharmacodynamics, one may expect to have improved tocolysis when two agents are combined. In vitro studies have demonstrated that simultaneous blockade of these different pathways could result in an additive or even synergistic effect capable of producing better uterine relaxation than induced by each drug alone. Accordingly, the use of multiple agent therapies has been suggested as a way forward in tocolytic search. In an observational study, combination therapy without serious side effects has been used in the management of PTL at extremely early gestations by Ingemarsson et al.3 However, this was not tested in structured human trials.

The objective of this study was to compare the tocolytic efficacy and safety of the combination of atosiban and nifedipine against the single agent, atosiban in the treatment of PTL.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of preterm labour
* Women with singleton pregnancies

Exclusion Criteria:

* Women with preterm prelabour rupture of membranes
* Women with any indication for emergency delivery for whom prolongation of pregnancy is contraindicated

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Participants will be followed for the duration of pregnancy, an expected average of 10 weeks
  Safety was assessed by maternal, fetal and neonatal adverse events. Particular emphasis was placed on serious adverse cardiovascular events, including cardiac arrest, respiratory arrest, admission to intensive care unit and death were assessed as serious maternal outcomes and perinatal complications were recorded by neonatal morbidity and mortality until discharge from the hospital
Number of women undelivered 48 hrs and seven days of initiation of therapy | Participants who are not delivered within seven days of initiation of therapy
  Tocolytic efficacy was assessed in terms of the proportion of women undelivered 48 hrs and seven days of initiation of therapy without the need for rescue tocolysis.
Number of Babies with Adverse Events as a Measure of Safety and Tolerability | participants will be followed for the duration of hospital stay, an expected average of 7 weeks
  Safety was assessed by maternal, fetal and neonatal adverse events. Perinatal complications were recorded by neonatal morbidity and mortality until discharge from the hospital

SECONDARY OUTCOMES:
Prolongation of pregnancy | Assessed till the date of delivery, an expected average of 10 weeks
Neonatal intensive care unit (NICU) admission | Till the time of discharge, an expected avearge of 7 weeks
  Number of neonates who are needing NICU admission after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Wafa R AlOmari, Principal Investigator — Tawam Hospital
Locations (2):
- United Arab Emirates (2):
  - Department of obstetrics and Gynecology, Tawam Hospital, Al Ain City, Abudhabi
  - Tawam Hospital, Al Ain City, Abudhabi

REFERENCES:
- [Background] Vogel JP, Nardin JM, Dowswell T, West HM, Oladapo OT. Combination of tocolytic agents for inhibiting preterm labour. Cochrane Database Syst Rev. 2014 Jul 11;2014(7):CD006169. doi: 10.1002/14651858.CD006169.pub2. PMID 25010869
- [Result] Doret M, Mellier G, Gaucherand P, Saade GR, Benchaib M, Frutoso J, Pasquier JC. The in vitro effect of dual combinations of ritodrine, nicardipine and atosiban on contractility of pregnant rat myometrium. BJOG. 2003 Aug;110(8):731-4. PMID 12892684
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046
- See also: RCOG Guidelines No.1 (B) February 2011. Tocolytic drugs for women in preterm labour. — http://rcog.org.uk